CLINICAL TRIAL: NCT04394130
Title: " Analgesic Efficacy of Continuous Infusion of Local Anaesthetic Versus Single-shot Injection Interscalene Brachial Plexus Block in Patients Receiving a Large Multimodal Analgesia: a Randomized Controlled Trial "
Brief Title: Analgesic Efficacy of Continuous Infusion of Local Anaesthetic Versus Single-shot Injection Interscalene Block
Acronym: BIGKIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Principal Investigator PD Dr Eric Albrecht, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00957
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Analgesia
Keywords: Regional anesthesia; Brachial plexus block; Shoulder surgery; Local anesthetics; Multimodal analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CI group (Experimental): Patients will have a preoperative ultrasound-guided interscalene brachial plexus block with 20 ml of lidocaïne 1% and epinephrine 1:100,000, followed by the insertion of a catheter. In the post-operative period, after clinical assessment of motor recovery in the operated limb (flexion of the forearm possible) in order to exclude any neurological damage of surgical origin, ropivacaine 0.5% 20 ml will be injected through the catheter.
  Then a continuous infusion of ropivacaine 0.2% at a flow rate of 6 ml.h-1 will be running for 48h after the bolus administration.
  During surgery, patients will also receive multimodal analgesia inclusive of iv dexamethasone 8 mg, iv magnesium sulfate 40 mg.kg-1, iv ketorolac 30 mg, and iv acetaminophen 1000 mg, according to the current practice in our institution.
  Interventions: Drug: ropivacaine 0.2%
- SS group (No Intervention): Patients will have a preoperative ultrasound-guided interscalene brachial plexus block with 20 ml of lidocaïne 1% and epinephrine 1:100,000, followed by the insertion of a catheter. In the post-operative period, after clinical assessment of motor recovery in the operated limb (flexion of the forearm possible) in order to exclude any neurological damage of surgical origin, ropivacaine 0.5% 20 ml will be injected through the catheter.
  After the injection, the catheter will be removed.
  During surgery, patients will also receive multimodal analgesia inclusive of iv dexamethasone 8 mg, iv magnesium sulfate 40 mg.kg-1, iv ketorolac 30 mg, and iv acetaminophen 1000 mg, according to the current practice in our institution.

INTERVENTIONS:
Drug: ropivacaine 0.2% — continuous peripheral nerve local anesthetic infusion (ropivacaïne 0.2 %) for 48 hours postoperative.
  Arms: CI group

SUMMARY:
The aim of this study is to study the analgesic efficacy of a continuous infusion of local anaesthetics for interscalene brachial plexus block after major shoulder surgery in the setting of multimodal analgesia, in order to determine whether the use of a catheter is still necessary in a contemporary practice.

DETAILED DESCRIPTION:
The hypothesis of this study is that in contemporary practice, comprising the administration of multimodal analgesia, the continuous infusion of local anesthetic via a catheter remains superior in terms of analgesia at 24 h compared to a single-shot injection at the level of the interscalene brachial plexus after major shoulder surgery.

This prospective randomized monocentric superiority study will include two parallel groups: a SS (single-shot injection) group and a CI (continuous infusion) group.

All patients will have a preoperative ultrasound-guided interscalene brachial plexus block with 20 ml of lidocaïne 1% and epinephrine 1:100,000, followed by the insertion of a catheter. In the post-operative period, after clinical assessment of motor recovery in the operated limb (flexion of the forearm possible) in order to exclude any neurological damage of surgical origin, ropivacaine 0.5% 20 ml will be injected through the catheter. In the SS group, the catheter will be removed. In the CI group, a continuous infusion of ropivacaine 0.2% at a flow rate of 6 ml.h-1 will be running for 48h after the bolus administration of ropivacaine 0.5%.

In both groups, patients will receive during surgery multimodal analgesia inclusive of iv dexamethasone 8 mg, iv magnesium sulfate 40 mg.kg-1, iv ketorolac 30 mg, and iv acetaminophen 1000 mg, according to the current practice in our institution.

Assignment to one of these two groups will be done according to a computer-generated list of random numbers, and the sealed envelopes method will be used.

In the postoperative period, patients will be prescribed an iv pca of morphine.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a major shoulder surgery (total shoulder arthroplasty or rotator cuff repair);
* ASA class 1 to 3;
* age more than 18 years old.

Exclusion Criteria:

* patient refusal or inability to understand and/or sign the inform consent
* contraindication for perineural block (allergy to local anesthetics, infection of puncture site, major coagulopathy, sensitive or motor deficiency on the operative side arm);
* chronic alcool abuse;
* chronic pain under chronic opioid treatment
* opioid drug abuse or under substitution treatment
* patients known for allergies to paracetamol, non steroidal anti inflammatory drugs, dexamethasone, sulfate magnesium, ondansetron, droperidol, and omeprazole;
* patients under chronic corticotherapy
* patients known for malignant hyperthermia;
* patients with chronic kidney failure class 3 or more;
* patients with severe pulmonary disease;
* patients with history of neck surgery or radiotherapy on the operative side;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
total i.v. morphine consumption | 24 hours postoperatively
  i.v morphine consumption in milligrams

SECONDARY OUTCOMES:
total i.v. morphine consumption postoperative | in the postoperative care unit, at 12 hours, 36 hours, and 48 hours postoperatively
  i.v morphine consumption in milligrams
pain scores at rest and on movement | in the postoperative care unit, and twice a day during the first 48 hours postoperatively
  Numeric pain intensity scale. Pain scores range from 0 (no pain) to 10 (worst possible pain).
presence of PONV | in the postoperative care unit and twice a day at 24 hours and 48 hours postoperatively
  verbal question to the patient if he has PONV or not
presence of pruritus | in the postoperative care unit and twice a day at 24 hours and 48 hours postoperatively
  verbal question to the patient if he has pruritus or not
overall patient satisfaction rate | at 24 hours and 48 hours postoperatively
  Numeric rating scale ranging from 0 (totally dissatisfied) to 10 (maximal satisfaction)
length of hospital stay | From operative day to hospital discharge or death during hospitalisation whichever came first, assessed up to 3 months
  in days
rate of complications related to the catheter | From operative day to hospital discharge or death during hospitalisation whichever came first, assessed up to 3 months
  infection at puncture point, catheter accidental removal
joint amplitude during anterior elevation of the shoulder | at 24 hours and 48 hours postoperatively
  Evaluated by physiotherapists
joint amplitude during shoulder abduction | at 24 hours and 48 hours postoperatively
  Evaluated by physiotherapists
joint amplitude during external rotation of the shoulder | at 24 hours and 48 hours postoperatively
  Evaluated by physiotherapists
pain score | at 3 months postoperatively
  Via phone contact. Numeric pain intensity scale. Pain scores range from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhyner P, Cachemaille M, Goetti P, Rossel JB, Boand M, Farron A, Albrecht E. Single-bolus injection of local anesthetic, with or without continuous infusion, for interscalene brachial plexus block in the setting of multimodal analgesia: a randomized controlled unblinded trial. Reg Anesth Pain Med. 2024 May 7;49(5):313-319. doi: 10.1136/rapm-2023-104681. PMID 37541683